CLINICAL TRIAL: NCT06106763
Title: The Effect Of Mandala Colouring On Anxiety, Depression, Pain And Quality of Life in Patients Receiving Haemodialysis Treatment
Brief Title: Mandala Colouring On Anxiety, Depression, Pain And Quality of Life
Acronym: MANDALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Ayşe Nefise BAHÇECİK, Prof., Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23.05.2022-2022/05
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hemodialysis Patients
Keywords: Hemodialysis; Anxiety; Depression; Pain; Quality of Life; Mandala painting
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Mandala and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala group (Experimental): Mandala coloring page
  Interventions: Other: Mandala coloring
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Mandala coloring — Mandala coloring page
  Other Names: Control group
  Arms: Mandala group

SUMMARY:
The research was conducted as an experimental research to determine the effect of mandala painting on pain, anxiety, depression and quality of life in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
The effect of mandala painting on pain, anxiety, depression and quality of life in patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

be over 18 Ability to communicate adequately Absence of psychiatric problems Volunteering to participate in the research Receiving hemodialysis treatment for at least 3 months

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analogue Scale (VAS) | 3. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Hospital Anxiety and Depression Scale (HAD) | 1. week
  The scale was designed to screen anxiety and depression mood states in the population with physical illness in a short time. The HAD scale consists of 2 subscales and 14 items scored between 0-3 as a 4-point Likert-type scale. The anxiety subscale includes items 1, 3, 5, 7, 9, 11 and 13 and is scored between 0-21, the depression subscale includes items 2, 4, 6, 8, 10, 12 and 14 and is scored between 0-21. The scoring of items 1, 3, 5, 6, 8, 10, 11 and 13 is 3,2,1,0, while the scoring of items 2, 4, 7, 9, 12 and 14 is 0,1,2,3. A score above 7 in the depression subscale is compatible with depression, while a score above 10 in the anxiety subscale is compatible with anxiety.
Hospital Anxiety and Depression Scale (HAD) | 3. week
  The scale was designed to screen anxiety and depression mood states in the population with physical illness in a short time. The HAD scale consists of 2 subscales and 14 items scored between 0-3 as a 4-point Likert-type scale. The anxiety subscale includes items 1, 3, 5, 7, 9, 11 and 13 and is scored between 0-21, the depression subscale includes items 2, 4, 6, 8, 10, 12 and 14 and is scored between 0-21. The scoring of items 1, 3, 5, 6, 8, 10, 11 and 13 is 3,2,1,0, while the scoring of items 2, 4, 7, 9, 12 and 14 is 0,1,2,3. A score above 7 in the depression subscale is compatible with depression, while a score above 10 in the anxiety subscale is compatible with anxiety.
Kidney Disease Quality of Life Form (KDQOL-36) | 1. week
  The first part of the KDQOL-36 (items 1-12) includes the medical outcomes study short form 12 health survey (SF-12) as a generic core. It includes questions about general health, activity limits, ability to accomplish desired tasks, depression and anxiety, energy level, and social activities. These 12 items make up the physical component summary (PCS) and mental component summary (MCS) scales. Some items contribute most to the PCS scale (items 1-5 and 8), whereas other items contribute most to the MCS scale (items 6, 7, and 9-12). The second part (items 13-16) constitutes burden of kidney disease subscale. It includes questions about how much kidney disease interferes with daily life, takes up time, causes frustration, or makes the respondent feel like a burden. The third part (items 17-28) covers symptoms and problem list subscale. It includes questions about how bothered a respondent feels by sore muscles, chest pain, cramps, itchy or dry skin, shortness of breath, faintness, lack o
Kidney Disease Quality of Life Form (KDQOL-36) | 3. week
  The first part of the KDQOL-36 (items 1-12) includes the medical outcomes study short form 12 health survey (SF-12) as a generic core. It includes questions about general health, activity limits, ability to accomplish desired tasks, depression and anxiety, energy level, and social activities. These 12 items make up the physical component summary (PCS) and mental component summary (MCS) scales. Some items contribute most to the PCS scale (items 1-5 and 8), whereas other items contribute most to the MCS scale (items 6, 7, and 9-12). The second part (items 13-16) constitutes burden of kidney disease subscale. It includes questions about how much kidney disease interferes with daily life, takes up time, causes frustration, or makes the respondent feel like a burden. The third part (items 17-28) covers symptoms and problem list subscale. It includes questions about how bothered a respondent feels by sore muscles, chest pain, cramps, itchy or dry skin, shortness of breath, faintness, lack o

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE NEFİSE BAHÇECİK, PhD, Study Director — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study should not be disclosed before publication

REFERENCES:
- [Background] Choi H, Hahm SC, Jeon YH, Han JW, Kim SY, Woo JM. The Effects of Mindfulness-Based Mandala Coloring, Made in Nature, on Chronic Widespread Musculoskeletal Pain: Randomized Trial. Healthcare (Basel). 2021 May 28;9(6):642. doi: 10.3390/healthcare9060642. PMID 34071674